CLINICAL TRIAL: NCT02302105
Title: Prospective Phase III Randomized Trial of Prostate Only or Whole Pelvic RadioTherapy in High Risk Prostate Cancer (POP-RT) Trial
Brief Title: Randomized Trial of Prostate Only or Pelvic RT in High Risk Prostate Cancer
Acronym: POP-RT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr Vedang Murthy, Dr Vedang Murthy, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP-RT
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate Only (Active Comparator): 66-68 Gray (Gy) in 25 fractions will be prescribed for the prostate PTV
  Interventions: Radiation: IGRT
- Whole Pelvis (Experimental): 66-68 Gray (Gy) in 25 fractions will be prescribed for the prostate PTV and 50 Gy in 25 fractions to nodal region .
  Interventions: Radiation: IGRT

INTERVENTIONS:
Radiation: IGRT — Image Guided RT to the prostate

SUMMARY:
Evidence to justify the use of the pelvic field is lacking for men with high risk localized prostate cancer. An additional randomized study is needed in men with a potential risk of nodal involvement to test the hypothesis that the use of the pelvic field contributed to the benefit observed in those studies.

This trial aims to compare the outcomes with whole pelvis RT and Prostate alone RT in patients with High risk, non metastatic Prostate cancer with a Lymph nodal >20% with Primary 5 year Biochemical failure free survival and Secondary Disease free survival, overall survival, Acute toxicity, Late toxicity and QOL Patients will be randomized to one of two arms Arm 1 Whole pelvis radiotherapy and Arm 2 Prostate only radiotherapy. The Dose prescription will be 66 Gy in 25 fractions will be prescribed for the prostate PTV in Arm 2 an additional 50 Gy in 25 fractions for nodal PTV in patients in Arm 1. An overlap volume at rectal-prostate interface will receive 64 Gy/25#.

All patients will receive hormone therapy starting at least 8 weeks prior to the beginning of radiotherapy. They will continue the hormone therapy and later for a total duration of 2-3 years.

ELIGIBILITY:
Inclusion

1. Any age according to the fitness estimated by the Physician
2. Physician estimated life expectancy > 5 years
3. Biopsy proven Adenocarcinoma of prostate
4. High risk prostate cancer based on Staging and Risk of Pelvic Nodal Metastases ≥ 20% as per the Roach formula (2/3 PSA) + [(GS - 6) x 10] If Gleason Score 8-10 - Any PSA, T1- T3a N0 M0 If Gleason Score 7 - PSA > 15, T1-T3a N0 M0 If Gleason Score 6 - PSA > 30, T1-T3a N0 M0 T3b-T4a N0 M0, Any Gleason Score, Any PSA
5. Ability to receive long term hormone therapy/ Orchidectomy
6. KPS ≥ 70 (see appendix)
7. Estimated life expectancy > 5 years
8. No previous history of malignancy ≤5 years
9. No prior history of therapeutic irradiation to pelvis
10. Patient willing and reliable for follow-up and QOL
11. No major co morbidities preventing radical treatment
12. Signed study specific consent form

Exclusion

1. Any histopathology other than Adenocarcinoma
2. Contraindication to Pelvic Radiotherapy like Inflammatory Bowel Disorders
3. No prior history of pelvic surgery
4. Uncontrolled diabetes
5. Uncontrolled cardiac co morbidity
6. Presence of nodal or distant metastatic disease

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2011-11-25 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Biochemical Disease Free Survival | 5 years
  Biochemical failure is defined using the standard Phoenix consensus definition i.e. PSA>2ng/ml over the nadir PSA

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Vedang Murthy, Navi Mumbai, Maharashtra, India

REFERENCES:
- [Result] Maitre P, Maheshwari G, Sarkar J, Singh P, Kannan S, Dutta S, Phurailatpam R, Raveendran V, Prakash G, Menon S, Joshi A, Pal M, Arora A, Murthy V. Late Urinary Toxicity and Quality of Life With Pelvic Radiation Therapy for High-Risk Prostate Cancer: Dose-Effect Relations in the POP-RT Randomized Phase 3 Trial. Int J Radiat Oncol Biol Phys. 2024 Oct 1;120(2):537-543. doi: 10.1016/j.ijrobp.2024.03.023. Epub 2024 Mar 28. PMID 38552989
- [Result] Murthy V, Maitre P, Kannan S, Panigrahi G, Krishnatry R, Bakshi G, Prakash G, Pal M, Menon S, Phurailatpam R, Mokal S, Chaurasiya D, Popat P, Sable N, Agarwal A, Rangarajan V, Joshi A, Noronha V, Prabhash K, Mahantshetty U. Prostate-Only Versus Whole-Pelvic Radiation Therapy in High-Risk and Very High-Risk Prostate Cancer (POP-RT): Outcomes From Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Apr 10;39(11):1234-1242. doi: 10.1200/JCO.20.03282. Epub 2021 Jan 26. PMID 33497252
- [Result] Murthy V, Maitre P, Bhatia J, Kannan S, Krishnatry R, Prakash G, Bakshi G, Pal M, Menon S, Mahantshetty U. Late toxicity and quality of life with prostate only or whole pelvic radiation therapy in high risk prostate cancer (POP-RT): A randomised trial. Radiother Oncol. 2020 Apr;145:71-80. doi: 10.1016/j.radonc.2019.12.006. Epub 2020 Jan 7. PMID 31923712